CLINICAL TRIAL: NCT05718830
Title: Selecting Specific Bio-markers and Researching Mechanisms of Immune Regulation From Inhalation Injury and Traumatic Lung Injury Based on Single Cell Sequencing Technology
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChiCTR2200056981
Record Dates: First submitted 2022-12-25; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Traumatic Lung Injury; Inhalation Injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with traumatic lung injury (TLI)
- patients with inhalation injury (ILI)
- health controls(HCs)

SUMMARY:
The goal of this observational study is to profile the circulating immunological traits of patients with traumatic lung injury (TLI) and inhalation injury (ILI),providing a new direction for the depth research of the pathogenesis, and providing new immune-related targets for diagnosis of the severity of lung injury and treatment.

The investigators performed scRNA-seq of neutrophil and peripheral blood mononuclear cells (PBMCs) from 10 ml fresh circulating blood from 3 patients with TLI and 3 patients with ILI at longitudinal timepoints,as well as peripheral blood from 3 health controls(HCs).

DETAILED DESCRIPTION:
The investigators performed single-cell transcriptomic sequencing (BD Rhapsody) on neutrophil and PBMCs extracted from the fresh circulating blood from 3 patients with TLI and 3 patients with ILI at longitudinal timepoints,as well as peripheral blood from 3 health controls(HCs). Three time points are picked by clinical conditions of patients with TLI or ILI: day 1 post hospital admission, day 3 post hospital and the day before discharged which matched to acute stage,progressive stage and convalescence.

ELIGIBILITY:
Inclusion Criteria:

1. Lung injury caused by burn trauma is confirmed, and the patient is hospitalized within 24 hours after burn or trauma (the clinician can make a definite diagnosis of lung injury based on the comprehensive judgment of the patient's etiology, history, clinical manifestations, blood gas analysis, laboratory tests and imaging);
2. Patients with inhalation injury caused by head, face and neck burns or inhalation injury combined with multiple body burns < 30%;
3. Patients with simple inhalation injury;
4. The normal control group should have no smoking history and be normal population;
5. According to the provisions of Good Clinical Practice(GCP), the informed consent has been obtained and the informed consent has been signed to volunteer for the test.

Exclusion Criteria:

1. Basic pulmonary diseases like chronic obstructive pulmonary disease (COPD), asthma and et al;
2. Severe organ dysfunction;
3. Autoimmune diseases;
4. Tumor;
5. Severe infection;
6. Pregnant or nursing women;
7. Fatal or life-threatening events caused by trauma;
8. Any history which may interfere the results or increase the risk of patients judged by researchers.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 patients with TLI and 3 patients with ILI age from 18 to 90 years old, admission within 24h after injury and diagnosed as traumatic lung injury by 2 surgeons on account of injury history and chest CT images. As well as peripheral blood from 3 health controls(HCs) who have no smoking history.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Computerized tomography, CT | 1day
  according to the proportion of rib fracture, pneumothorax, hemothorax,lung contusion in the image
Computerized tomography, CT | 3 day
  according to the proportion of rib fracture, pneumothorax, hemothorax,lung contusion in the image
Computerized tomography, CT | through study completion, an average of 2 weeks
  according to the proportion of rib fracture, pneumothorax, hemothorax,lung contusion in the image
Partial pressure of carbon dioxide in arterial blood, PaCO2 | 1day
Partial pressure of carbon dioxide in arterial blood, PaCO2 | 3 day
Partial pressure of carbon dioxide in arterial blood, PaCO2 | through study completion, an average of 2 weeks
Oxygenation index and Fraction of Inspired Oxygen will be combined to report FiO2/PaO2 | 1 day
Oxygenation index and Fraction of Inspired Oxygen will be combined to report FiO2/PaO2 | 3 day
Oxygenation index and Fraction of Inspired Oxygen will be combined to report FiO2/PaO2 | through study completion, an average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Burn Surgery, the First Affiliated Hospital of Naval Medical University, Shanghai, Shanghai Municipality, China